CLINICAL TRIAL: NCT05609110
Title: Safety and Efficacy of Remote Ischemic Conditioning for Spontaneous Intracerebral Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SERIC-ICH
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Intracranial Hemorrhages
Keywords: Intracranial Hemorrhage; remote ischemic conditioning
MeSH Terms: conditions — Intracranial Hemorrhages

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Active Comparator): Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 200 mmHg.
  Interventions: Device: Remote ischemic conditioning
- Sham RIC group (Placebo Comparator): Sham remote ischemic conditioning (Sham RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mm Hg.
  Interventions: Device: Sham remote ischemic conditioning

INTERVENTIONS:
Device: Remote ischemic conditioning — Remote ischemic conditioning is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 200 mmHg.
  Arms: RIC group
Device: Sham remote ischemic conditioning — Remote ischemic conditioning is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 60 mmHg.
  Arms: Sham RIC group

SUMMARY:
The purpose of this study is to determine the efficacy and safety of remote ischemic conditioning in treating acute intracerebral hemorrhage.

DETAILED DESCRIPTION:
Spontaneous intracerebral hemorrhage is a major cause of disability and mortality among different types of stroke, and few effective treatment options are available. Therefore, it is essential to develop new approaches to improve the prognosis of these patients. Recently, remote ischemic conditioning (RIC), a method that involves inducing multiple brief episodes of ischemia and reperfusion in the limbs, has been indicated to exert neuroprotective effects in experimental stroke. The underlying neuroprotective mechanism triggered by RIC induces gene expression, alters pathways, promotes neurogenesis and blood vessel development, reduces oxidative stress and neuronal apoptosis, and inhibits proinflammatory signals. Previously, several clinical trials have shown that single or repeated RIC treatments for cerebrovascular diseases are feasible and safe. Therefore, we hypothesize that RIC could improve functional outcome in patients with intracerebral hemorrhage. We design this prospective, multicenter, randomized controlled trial to evaluate the efficacy and safety of RIC in treating intracerebral hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Supratentorial intracerebral hemorrhage confirmed by brain CT scan.
3. No disability in the community before ICH (premorbid mRS≤ 1).
4. NIHSS score ≥ 6 and GCS ≥ 8 upon presentation.
5. Able to commence RIC treatment within 24 hours of stroke onset.
6. Systolic blood pressure ≤ 180 mmHg before randomization.
7. Signed and dated informed consent is obtained.

Exclusion Criteria:

1. Definite evidence of secondary ICH, such as structural abnormality, brain aneurysm, brain tumor, thrombolytic drug.
2. Hematoma with a mid-line shift, cerebral herniation or isolate intraventricular hemorrhage.
3. Already booked for surgical treatment.
4. Life expectancy of less than 180 days due to comorbid conditions.
5. Concurrent use of anticoagulation drugs including Warfarin, dabigatran, rivaroxaban or coagulopathy (defined as INR, APTT, and PT beyond the upper limit of normal range).
6. Any soft tissue, orthopedic, or vascular injury, wounds or fractures in healthy upper limb which may pose a contraindication for application of RIC.
7. Severe hepatic and renal dysfunction, or ALT/AST >3 times upper limit of normal, or serum creatinine >265umol/l.
8. Known pregnancy or breastfeeding.
9. Patients being enrolled or having been enrolled in other clinical trial within 3 months prior to this clinical trial.
10. A high likelihood that the patient will not adhere to the study treatment and follow up regimen.
11. Patients unsuitable for enrollment in the clinical trial according to investigators decision making.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Modified Rankin Scale (mRS) Score 0-2 at 180 days | 180 days
  Proportion of patients with Modified Rankin Scale (mRS) Score 0-2. Ranged from 0 to 6, a low value represents a better outcome.

SECONDARY OUTCOMES:
Proportion of patients with Modified Rankin Scale (mRS) Score 0-2 at 90 days | 90 days
  Proportion of patients with Modified Rankin Scale (mRS) Score 0-2. Ranged from 0 to 6, a low value represents a better outcome.
Ordinal shift of the full range of mRS scores at 90 and 180 days | 90 days, 180 days
  Ranged from 0 to 6, a low value represents a better outcome.
Hematoma growth at 24 hours | 24 hours
  The growth in hematoma volume after the onset of intracerebral hemorrhage, which is assessed by Computed Tomography (CT) brain scan.
National Institute of Health stroke scale (NIHSS) at 7 days | 7 days
  National Institute of Health stroke scale (NIHSS) ranged from 0 to 42, a low value represents a better outcome.
Adverse events occurring in the course of the study. | 6 months
  The safety endpoints will include all adverse events, severe adverse events and RIC related adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China